CLINICAL TRIAL: NCT01198275
Title: N-3 Polyunsaturated Fatty Acids (n-3 PUFAs) in the Prevention of Atrial Fibrillation Recurrences After Electrical Cardioversion. A Prospective Randomized Study.
Brief Title: n-3 Polyunsaturated Fatty Acids (PUFAs) in the Prevention of Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Savina Nodari, N-3 Polyunsaturated Fatty Acids (n-3 PUFAs) in the Prevention of Atrial Fibrillation Recurrences After Electrical Cardioversion. A Prospective Randomized Study., Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS-PUFA-01
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Atrial Fibrillation
Keywords: PUFA atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Omacor; Amiodarone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- n-3 PUFAs (Active Comparator)
  Interventions: Drug: n-3 PUFAs; Drug: RASS inhibitors and/or RAS blockers; Drug: Amiodarone
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: RASS inhibitors and/or RAS blockers; Drug: Amiodarone

INTERVENTIONS:
Drug: n-3 PUFAs — 1.0 g of EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) in the average ratio EPA/DHA of 0.19:1.5, one capsule twice a day
  Other Names: OMACOR
  Arms: n-3 PUFAs
Drug: Placebo — 1.0 g of olive oil,one capsule twice a day
  Arms: placebo
Drug: RASS inhibitors and/or RAS blockers — Patients on ACE-Is or ARBs were continued on the same agent. In those who were not on therapy, an ACE-I or an ARB was started. In all patients, an effort was made to achieve the highest tolerated dose.
  Other Names: renin-angiotensin-aldosterone system inhibitor
Drug: Amiodarone — Patients on amiodarone were continued at a maintenance dose of 200 mg daily, whereas those who were not taking amiodarone were started at a dose of 400 mg daily for 1 week and then continued on a maintenance dose of 200 mg daily.

SUMMARY:
The purpose of this study is to determine the effect of n-3 PUFAs in addition to amiodarone and renin-angiotensin-aldosterone system (RAAS) inhibitors on the maintenance of sinus rhythm after electrical conversion in patients with persistent Atrial fibrillation (AF).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia and represents an increasing burden on the healthcare system. Treatment of AF remains controversial. In patients on antiarrhythmic therapy, the one-year relapse rates of AF after cardioversion ranges from 44% to 77% at one year and amiodarone appears to the be the most effective in maintaining sinus rhythm.Over the last few years, a growing amount of evidences has supported the protective effects of n-3 PUFAs in preventing ventricular arrhythmias and reducing the risk of sudden cardiac death. Furthermore, in the last years, the interest for their possible beneficial role in AF prevention has been increasing.We hypothesized that the administration of n-3 PUFAs could reduce the AF recurrence rate more than amiodarone plus RAAS inhibitors in patients with persistent AF. Therefore the present study aims to evaluate the role of n-3 PUFAs in the prophylaxis of AF recurrences after DCCV in addition to amiodarone and RAS blockers therapy in patients with persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* persistent Atrial Fibrillation (AF) lasting > one month
* history of at least one AF relapse after previous electrical or Pharmacological cardioversion

Exclusion Criteria:

* left atrium size > 6 cm
* severe valvulopathy
* myocardial infarction during the previous 6 months
* unstable angina
* NYHA heart failure class IV or hemodynamic instability
* cardiac surgery during the previous 3 months
* significant pulmonary thyroid and hepatic disease
* contraindications to treatment with amiodarone or RASS inhibitors
* chronic renal dysfunction
* QT > 480 msec in the absence of bundle-branch block
* bradycardia < 50 b/min
* diagnosis of paroxysmal AF
* hyperkalemia
* pregnancy
* any disease or other medical treatment that, in the opinion of the investigators, could interfere with the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Savina Nodari, MD, Principal Investigator — Department of Experimental and Applied Medicine-Section of Cardiovascular Diseases; Livio Dei Cas, MD, Study Director — Department of Experimental and Applied Medicine-Section of Cardiovascular Diseases
Locations (1):
- Arrhytmias and Heart failure Unit-Spedali Civili Hospital, Brescia, Brescia, Italy

REFERENCES:
- [Background] 1) Go AS, Hylek EM. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA 285(18):2370-2375, 2001 2) Wolf PA, Mitchell JB. Impact of atrial fibrillation on mortality, stroke, and medical costs. Arch Intern Med.;158(3):229-234, 1998 3) de Denus S, Sanoski CA. Rate vs rhythm control in patients with atrial fibrillation: a meta-analysis. Arch Intern Med 165(3):258-262, 1998 4) Fuster V, Ryden LE. ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation.Europace 8(9):651-745, 2006 5) Nichol G, McAlister F. Meta-analysis of randomised controlled trials of the effectiveness of antiarrhythmic agents at promoting sinus rhythm in patients with atrial fibrillation. Heart 87(6):535-543, 2002 6) Calo L, Bianconi L. N-3 Fatty acids for the prevention of atrial fibrillation after coronary artery bypass surgery: a randomized, controlled trial. J Am Coll Cardiol 45(10):1723-1728, 2005
- [Derived] Nodari S, Triggiani M, Campia U, Manerba A, Milesi G, Cesana BM, Gheorghiade M, Dei Cas L. n-3 polyunsaturated fatty acids in the prevention of atrial fibrillation recurrences after electrical cardioversion: a prospective, randomized study. Circulation. 2011 Sep 6;124(10):1100-6. doi: 10.1161/CIRCULATIONAHA.111.022194. Epub 2011 Aug 15. PMID 21844082
- See also: interview during American College of Cardiology 2010 convention — http://www.theheart.org

RESULTS

PARTICIPANT FLOW:
Groups:
- n-3 PUFAs: 1.0 g gelatin capsules containing a total of 850 mg to 882 mg of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) ethyl esters with an average ratio EPA/DHA of 0.9:1.5 twice daily
- Placebo: 1.0 g placebo gelatine capsules(olive oil)twice daily
Period: Overall Study
Arm/Group | n-3 PUFAs | Placebo
Started | 100 | 99
Completed | 94 | 94
Not Completed | 6 | 5
Not completed — Adverse Event | 2 | 3
Not completed — spontaneous return to sinus rhythm | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | n-3 PUFAs | Placebo | Total
Number analyzed (Participants) | 100 | 99 | 199
Age Continuous [Mean (Standard Deviation); unit: years] | 70 (6) | 69 (9) | 69.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 36 | 66
  Male | 70 | 63 | 133

OUTCOME MEASURES:

1. Secondary Outcome: The Mean Time to a First Recurrence of AF and the Rate of AF Recurrence
Description: The mean time to a first recurrence of AF; and the rate of AF recurrence at 1, 3 and 6 months.
Time Frame: 1, 3 and 6 months
Reporting Status: Not Posted, anticipated posting 2011-07
Measure: Mean (Standard Deviation); unit: time

2. Primary Outcome: Probability of Maintenance of Sinus Rhythm at One-year Follow up.(Number of Patients Who Maintained Sinus Rhythm)
Description: Sinus Rhythm maintenance means no Atrial Fibrillation recurrence at one-year follow up. Patients with successful electrical cardioversion (DCCV)underwent weekly clinical and electrocardiographic controls for the first three weeks following cardioversion. Subsequently, follow up visits with performance of clinical evaluation, ECG, and a 24-hour Holter monitoring were performed at 1, 3, 6 and 12 months after DCCV.
Time Frame: one year
Measure: Number; unit: partecipants
Arm/Group | n-3 PUFAs | Placebo
Number analyzed (Participants) | 100 | 99
partecipants | 61 | 34
Statistical Analysis 1: Comparison: n-3 PUFAs vs Placebo; Give a relapse rate ranging from 40% to 60% on ACE-I/ARB and amiodarone therapy, considering the high risk of relapses in our study population we conservatively assumed a 50% relapse rate. We calculated that a total of 180 patients would yield 80% power to detect a clinically relevant difference of about 20% in AF recurrence with the addition of n-3 PUFAs at a log-rank test, with a significance level of 0.05; Test type: Superiority or Other; p < 0.05, Kaplan Meyer analysis; The time to first AF recurrence was analyzed with the Kaplan-Meier method and compared with the log-rank test; Hazard Ratio (HR) = 0.441, 95% CI 2-sided [0.292 to 0.666] — Hazard ratios between n-3 PUFA and Placebo together with confidence intervals were estimated using the Cox proportional regression model

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | n-3 PUFAs | Placebo
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 0/100 | 0/99

LIMITATIONS AND CAVEATS:
The effect of n-3 PUFAs on the recurrence of Atrial Fibrillation (AF) in patients with persistent AF not on amiodarone and a renin-angiotensin-aldosterone system (RASS) inhibitor cannot be inferred from our findings

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No